CLINICAL TRIAL: NCT05102123
Title: PeRiopEratiVE SmokiNg CessaTion Trial
Acronym: PREVENT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022_09_01
Record Dates: First submitted 2021-10-19; First posted 2021-11-01 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Smoking (Tobacco) Addiction; Smoking Cessation
MeSH Terms: conditions — Smoking; Behavior, Addictive; Smoking Cessation | interventions — cytisine

STUDY DESIGN:
Intervention Model Description: 2x2 factorial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cytisine and Video Messaging (Experimental): Administration of cytisine (pharmaceutical support) to patients on a set dose schedule with behavioural support through video messaging.
  Interventions: Drug: Cytisine; Behavioral: Video Messaging
- Placebo and Video Messaging (Placebo Comparator): Administration of placebo (inactive drug) to patients on a set dose schedule with behavioural support through video messaging.
  Interventions: Behavioral: Video Messaging
- Cytisine and No Video Messaging (Active Comparator): Administration of cytisine (pharmaceutical support) to patients on a set dose schedule with behavioural support according to standard care such as a phone number for a self-help line.
  Interventions: Drug: Cytisine
- Placebo and No Video Messaging (No Intervention): Administration of placebo (inactive drug) to patients on a set dose schedule behavioural support according to standard care such as a phone number for a self-help line.

INTERVENTIONS:
Drug: Cytisine — Listed as a natural health product in Canada, cytisine is utilized to aid in smoking cessation
  Arms: Cytisine and No Video Messaging; Cytisine and Video Messaging
Behavioral: Video Messaging — Supportive messaging utilizing a video messaging platform to encourage patients to abstain from smoking throughout the treatment period.
  Arms: Cytisine and Video Messaging; Placebo and Video Messaging

SUMMARY:
PREVENT is a multicentre, 2x2 factorial, randomized clinical trial that aims to determine the effect of cytisine versus placebo, as well as the effect of video messaging to support smoking cessation versus standard of care in perioperative patients. This trial aims to investigate the effects of cytisine and text messaging on 6-month continuous abstinence rates. PREVENT will also assess secondary outcomes at 30 days, 56 days and 6 months post-randomization: 7-day point prevalence abstinence, urge to smoke, time to first lapse, time to relapse, number of cigarettes smoking if still smoking, pulmonary complications, vascular complications, wound and infectious complications, stroke, time in hospital and acute hospital care.

ELIGIBILITY:
Inclusion Criteria:

1. are ≥18 years of age
2. are scheduled to undergo surgery within 28 days
3. are a current smoker and not currently using any smoking cessation treatment and,
4. have a smart mobile phone with an active, up to date data plan and with internet access
5. provide informed consent to participate.

Exclusion Criteria:

1. are pregnant or breastfeeding or expecting to become pregnant during the study follow-up period
2. are deemed unreliable for study procedures or follow-up
3. have a documented allergic reaction to cytisine, or its components (non-medicinal ingredients) or to the non-medicinal ingredients of the placebo.
4. had myocardial infarction, unstable angina, or stroke/transient ischemic attack within the preceding 2 weeks.
5. will have surgery with expected nil intake by mouth for 2 or more days
6. have previously participated in PREVENT
7. have a known diagnosis of untreated pheochromocytoma; Schizophrenia/bipolar psychiatric illness and currently psychotic; currently having suicidal ideation or risk of suicide as determined by the site physician, known history of moderate to severe depression; currently uncontrolled severe hypertension (≥180/120 mmHg) despite treatment; known history of uncontrolled hyperthyroidism (thyrotoxicosis), severe renal impairment i.e., creatinine clearance of less than 30 ml per minute (Cockcroft- Gault equation) or receiving long-term dialysis, or known diagnosis of severe liver disease as determined by the site physician or documented in the clinical history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1720 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Smoking Cessation | 6 months
  complete abstinence (smoking not more than 5 cigarettes) beginning on day 5 post randomization and lasting until the assessment at 6 months post-randomization with biochemical verification for those who report abstinence, using exhaled breath carbon monoxide (cut-off <10 parts per million [ppm]) measured with a carbon monoxide (CO) monitor

SECONDARY OUTCOMES:
7-day point-prevalence abstinence at 30 days | 30 days
  Self-report of not smoking cigarettes [not even a puff] in the 7 days before the 30-day follow-up
7-day point-prevalence abstinence at 56 days | 56-days
  Self-report of not smoking cigarettes [not even a puff] in the 7 days before the 56-day follow-up
7-day point-prevalence abstinence at 6-months | 6-months
  Self-report of not smoking cigarettes [not even a puff] in the 7 days before the 6-month follow-up
Urge to smoke | baseline and 6-months
  urge to smoke using the Mood and Physical Symptoms Scale [MPSS] at baseline and 6 months; a higher score indicates a stronger urge to smoke; To assess the effect of abstinence calculate the change from baseline (just prior to stopping smoking) to the post-abstinence follow-up point for items 1 to 7 and 10 to 12, and take the raw scores for items 8 and 9
Number of cigarettes smoked daily if still smoking | 30 days, 56 days and 6 months
  Number of cigarettes smoked daily if still smoking
Time to first lapse | 6 months
  Time to first cigarette smoked after the initial quit, even a single puff
Time to relapse | 6 months
  Time to return to regular smoking for three or more concurrent days after a period of abstinence.
6 month continuous abstinence rate | 6-months
  Complete abstinence (smoking not more than 5 cigarettes) beginning on the quit date and lasting until the assessment at 6 months post-randomization with biochemical verification for those who report abstinence, using exhaled breath carbon monoxide (cut-off <10 ppm) measured with a carbon monoxide (CO) monitor.
  *Cigarettes smoked within 5 days of randomization will be discounted.
Wound complications | 6 months
  Seroma- wound drainage or repeated dressings required; Wound dehiscence or delayed wound healing
Infectious complications | 6 months
  Infection - defined as a pathologic process caused by the invasion of normally sterile tissue, fluid, or body cavity by pathogenic or potentially pathogenic organisms.
  Surgical site infection- An infection that occurs within 30 days after surgery and involves the skin, subcutaneous tissue of the incision (superficial incisional), or the deep soft tissue (e.g., fascia, muscle) of the incision (deep incisional).
  Sepsis- Based on the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). Sepsis requires a quick Sequential Organ Failure Assessment (qSOFA) Score ≥2 points due to infection. The qSOFA includes the following items and scoring system: 1. altered mental status (1 point); 2. systolic blood pressure ≤100 mm Hg (1 point); and 3. respiratory rate ≥22 breaths per minute (1 point).
Respiratory complications | 6 months
  Pneumonia - defined as an acute infection of the pulmonary parenchyma that is associated with at least one sign or symptom of lower respiratory acute infection (e.g., cough, pleuritic chest pain) or acute systemic illness (e.g., fever, chills, confusion, hypoxemia); accompanied by the presence of an acute infiltrate/consolidation on a chest radiograph or auscultatory findings consistent with pneumonia (such as crackles and/or localized rales) for which there is no other explanation.
  Respiratory insufficiency requiring ventilatory support - Patient intubated or put on bilevel positive airway pressure (BiPAP).
Non-fatal Myocardial infarction | 6 months
  according to the 4th universal definition
Number of Patients with Proximal venous thrombo-embolism | 6 months
  The diagnosis of PE requires any one of the following:
  1. A high probability ventilation/perfusion lung scan,
  2. An intraluminal filling defect of a segmental or larger artery on a helical computerized tomography (CT) scan,
  3. An intraluminal filling defect on pulmonary angiography, or
  4. A positive diagnostic test for deep venous thrombosis A. Non-diagnostic ventilation/perfusion lung scan B. Non-diagnostic helical CT scan.
  The diagnosis of proximal DVT (leg or arm) requires:
  1. Thrombosis involving the popliteal vein or more proximal veins for leg DVT and axillary or more proximal veins for arm DVT, AND
  2. Evidence of vein thrombosis by any one of the following:
  1. A persistent intraluminal filling defect on contrast venography, 2. Non-compressibility of one or more venous segments on B mode compression ultrasonography, or 3. A clearly defined intraluminal filling defect on contrast enhanced computed tomography.
Stroke | 6 months
  Stroke is defined as either: 1. a new focal neurological deficit thought to be vascular in origin with signs or symptoms lasting ≥24 hours or leading to death; or 2. a new focal neurological deficit thought to be vascular in origin with signs or symptoms lasting <24 hours with positive neuroimaging consistent with a stroke.
Non-fatal cardiac arrest | 6 months
  Nonfatal cardiac arrest is defined as successful resuscitation from either documented or presumed ventricular fibrillation, sustained ventricular tachycardia, asystole, or pulseless electrical activity requiring cardiopulmonary resuscitation, pharmacological therapy, or cardiac defibrillation.
Death | 6 months
  The definition of death is all cause mortality.
Length of hospital stay | time of hospital admission to time of discharge for surgical stay
  Defined as time of hospital admission to time of discharge from hospital after index surgery.
Acute hospital care since discharge | after hospital discharge for the study surgery to 6-month follow-up
  Acute-hospital care is a composite outcome of hospital re-admission (patient admission to an acute-care hospital) and emergency department visit (patient visit to an emergency department, which includes urgent-care centre visit).

OTHER OUTCOMES:
Health services utilization-related costs | 6-months
  Data on hospital re-admission, healthcare utilization, and costs of health service utilization will be obtained from the Institute for Clinical Evaluative Sciences data repository. Administrative databases used to describe the health service utilization include: 1. Registered Persons Database - demographics and vital statistics of all legal residents of Ontario; 2. Discharge Abstract Database - records of inpatient hospitalizations from the Canadian Institute for Health Information (CIHI); 3. Ontario Health Insurance Plan Database - physician billing claims, and the National Ambulatory Care Reporting System - information on emergency department visits from CIHI.
Health-related quality of life (HRQoL) | baseline and 6-months
  HRQoL will be measured with the EQ-5D-5L instrument (https://euroqol.org/eq-5d-instruments/sample-demo) due to its increased sensitivity and validation in several countries including Canada. The EQ-5D-5L is also recommended in Canada to calculate the Quality Adjusted Life Years (QALYs) when conducting cost-effectiveness analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Ofori, Dr., Principal Investigator — Population Health Research Institute; Flavia Kessler Borges, Dr., Principal Investigator — Population Health Research Institute
Locations (4):
- Canada (4):
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Kingston Health Science Centre with its research institute Kingston General Health Research Institute, Kingston, Ontario
  - Lawson Health Research Institute: London Health Sciences Centre Research Inc. and the Lawson Research Institute, London, Ontario

IPD SHARING:
Plan to Share IPD: No
The Population Health Research Institute (PHRI) is the sponsor of this trial. The PHRI believes the dissemination of clinical research results is vital and sharing of data is important. PHRI prioritizes access to data analyses to researchers who have worked on the trial for a significant duration, have played substantial roles, and have participated in raising the funds to conduct the trial. PHRI balances the length of the research study, and the intellectual and financial investments that made it possible with the need to allow wider access to the data collected. Data will be disclosed only upon request and approval of the proposed use of the data by a Review Committee.